CLINICAL TRIAL: NCT03974438
Title: Acupuncture (Dry-needling) as Treatment of Post-herpetic Neuralgia: A Double-blinded Randomized Clinical Trial.
Brief Title: Acupuncture as Treatment of Post-herpetic Neuralgia: A RCT A Double-blinded Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Martin Sollie, Principal investigator, M.D, Dept. of Plastic and Reconstructive Surgery Affiliation: Odense University Hospital Collaborators:, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S-20190101
Record Dates: First submitted 2019-06-01; First posted 2019-06-05 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Post Herpetic Neuralgia
Keywords: post-herpetic neuralgia; pain; post herpetic neuralgia; shingles; autologous fat grafting; autologous fat transplant
MeSH Terms: conditions — Neuralgia, Postherpetic; Pain; Herpes Zoster

STUDY DESIGN:
Intervention Model Description: The participants will be divided into two groups, group A, the intervention group, will receive SDN in the area of pain. Group B, the control group will receive a sham procedure.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will not be aware of the treatment given. The randomization will take place right before the procedure begins. The treatment will be given to the skin covering the spine and the patients will be placed in the supine position. They will therefore not know whether or not they are receiving the actual acupuncture or the sham procedure.
  The investigator will not be present at the procedures and will not have access to patients records and data until after the trial is complete.
  The outcomes are measured using validated questionnaires. They will be assessed by the investigator at the time of project completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Acupunture (SDN) (Experimental): Patients allocated to the intervention arm will receive SDN to the area of skin over the spine on the level of the specific dermatome involved in their chronic pain.
  Interventions: Procedure: Superficial dry needling / Acupunture
- Control - Sham acupunture (Sham Comparator): Patients allocated to the control arm will receive sham-SDN to the area of skin over the spine on the level of the specific dermatome involved in their chronic pain. The sham procedure consists of a blunted needle, that does not penetrate the skin.
  Interventions: Procedure: Superficial dry needling / Acupunture

INTERVENTIONS:
Procedure: Superficial dry needling / Acupunture — Se arm-description.

SUMMARY:
The aim of this study is to perform the first RCT investigating the possible effect of superficial dry-needling (SDN) - a special kind of acupuncture used for PHN. The participants will be divided into two groups. Group A, the intervention group will receive SDN in the area of pain. Group B, the control group will receive a sham procedure.

DETAILED DESCRIPTION:
The aim of this study is to investigate the possible effect of SDN on PHN. The study population consists of patients with chronic pain after herpes zoster.

The study is a controlled double-blinded randomized study. The participants will be divided into two groups, group A, the intervention group, will receive SDN in the area of pain. Group B, the control group will receive a sham procedure. The procedure will take place at the out-patient clinic at Odense University Hospital. The plan is to include 40 patients (20 in each group).

ELIGIBILITY:
Inclusion Criteria:

* Age between 50-75 years.
* Pain in the dermatomal area of the previous outbreak of HZ.
* Pain located to a dermatome originating from the thoracic or lumbar spine.
* At least six months since the outbreak.
* Understands the purpose of the study and is able to give consent.

Exclusion Criteria:

* A psychiatric illness affecting participation in the study.
* Active cancer
* Pregnancy

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Dermal pain [LEVEL OF PAIN] | 1 month
  Questionnaire. Visual Analogue Scale (VAS). Patients will be asked to report on their average and maximum level of pain on a scale from 0-10.

SECONDARY OUTCOMES:
Neuropathic pain [LEVEL OF PAIN] | 1 month
  Neuropathic Pain Symptom inventory (NPSI), Questionnaire. NPSI consists of 12 items in total: 10 items investigates differential symptoms descriptors and 2 items evaluate spontaneous and paroxysmal spontaneous pain.
  The tool evaluates mean pain intensity in the last 24h in a verbal numeric scale from zero (no pain) to 10 (worst imaginable pain). Total pain intensity score may be calculated by the sum of the 10 descriptors.
  The descriptors are:
  Burning, Squeezing, Pressure, Electric Shocks, Stabbing, Provoked by brushing. Provoked by pressure, Evoked by cold stimulation, Pins and needles, Tingling.
Quality of life [QUALITY OF LIFE/ SATISFACTION] | 1 month
  Short Form 36 (SF-36), Questionnaire. Scoring the RAND 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per a scoring key. All items are scored so that a high score defines a more favorable health state. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. After this, items in the same scale are averaged together to create the 8 scale scores.
  The eight health concepts are: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No